CLINICAL TRIAL: NCT02396628
Title: Multicentre Phase 2 Trial to Evaluate the Efficacy of Ruxolitinib in Steroid-refractory Acute Multicenter, Randomized Phase 2 Trial to Determine the Response Rate of Ruxolitinib and Best Available Treatment (BAT) Versus BAT in Steroid-refractory Acute Graft-versus-Host Disease (aGvHD)
Brief Title: Ruxolitinib In GvHD
Acronym: RIG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: impossibility to recruit in the BAT arm
Sponsor: Prof. Dr. Nikolas von Bubnoff (Other)
Collaborators: Clinical Trials Unit Freiburg (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Nikolas von Bubnoff, Coordinating Investigator, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIG-P000814; 2014-004267-20 (EudraCT Number); DRKS00007939 (Registry Identifier: DRKS)
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Graft vs Host Disease
Keywords: Graft-versus-Host Disease (GvHD); resistance to therapy; allogeneic stem cell transplantation; Ruxolitinib
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Treatment with Ruxolitinib at a dose of 10 mg BID orally addition to BAT according DGHO-Onkopedia guidelines.
  Interventions: Drug: Experimental intervention
- Standard treatment (Active Comparator): Treatment according to DGHO-Onkopedia guidelines for treatment of acute GvHD (as of March 2018). Optional cross over from BAT to Ruxolitinib and BAT in case of lack of response from day 28.
  Interventions: Drug: Standard treatment

INTERVENTIONS:
Drug: Experimental intervention — Treatment with Ruxolitinib at a dose of 10 mg BID orally addition to BAT according DGHO-Onkopedia guidelines
  Arms: Experimental intervention
Drug: Standard treatment — Treatment according to DGHO-Onkopedia guidelines for treatment of acute GvHD (as of March 2018). Optional cross over from BAT to Ruxolitinib and BAT in case of lack of response from day 28.
  Arms: Standard treatment

SUMMARY:
The preliminary data demonstrate potent activity of Ruxolitinib in steroid-refractory aGvHD. In this phase 2 trial the efficacy of Ruxolitinib and best available treatment (BAT) versus BAT in steroid-refractory acute GvHD in approximately 12 transplantation centers in Germany will be compared. The response by monitoring the clinical GvHD grade, requirement of alternative GvHD active agents and serum levels of pro-inflammatory cytokines will be determined.

DETAILED DESCRIPTION:
The pathophysiological hallmark of GvHD after allo-HCT is an allogeneic donor T cell re-sponse against recipient antigens. This process is aggravated by increased processing and presentation of host antigens by donor APCs following conditioning treatment. The al-logeneic T cell response leads to inflammation, tissue damage and fibrosis and is mediated by extensive production of inflammatory cytokines such as IL-1, IL-2R, IL-6 and TNF. The signal transmission of inflammatory cytokines in effector cells requires activation of specialized kinases from the family of the Janus kinases. These kinases, JAK1, 2 and 3 are linked to cytokine receptors, and are activated upon binding of the cytokine to the receptor of the inflammatory effector. The JAK1/2 kinase inhibitor Ruxolitinib (INC424) is approved for myelofibrosis. In advanced myelofibrosis, Ruxolitinib lead to sustained clinical remissions with regard to constitutional symptoms, weight loss and spleen size in the majority of treated patients. Of note, clinical responses correlated with a marked reduction in inflammatory plasma cytokines.

Importantly, cytokines down-regulated by Ruxolitinib in patients with myelofibrosis correspond to inflammatory effectors that mediate tissue damage and inflammation in GvHD. These are mainly the cytokines IL- 1, IL -6, TNF and IFN-gamma. Since Ruxolitinib suppresses the JAK1 / 2 cytokine response, we hypothesized that Ruxolitinib might attenuate the cytokine mediated inflammatory tissue damage in GVHD and thus might favourably affect the severity and course of GvHD after allo-HCT.

In vitro, we demonstrated in an allogeneic system (major mismatch mixed-lymphocyte reactions) that co-incubation with Ruxolitinib strongly suppressed both the proliferation of alloge-neic T cells and the production of inflammatory cytokines. Using a very aggressive major mismatch mouse model of acute GvHD Ruxolitinib treatment signifi-cantly prolonged survival of animals (see Figure 1A). In addition, in these animals showed a reduced weight loss, significantly reduced histopathological GvHD severity, suppression of inflammatory cytokines in the serum and a reduction of donor T cells in GvHD target organs such as the intestines.

Sole suppression of cytokine production or cytokine receptor activity by Ruxolitinib would be very similar to already established drugs for GvHD and no major conceptual advance. However we observed that Ruxolitinib did not only suppress cytokine production but also led to increased frequencies of FoxP3+ regulatory T cells. This cell type was previ-ously shown to lead to long-lasting tolerance as compared to the short-term immunosuppression achieved by conventional medication for GvHD.

ELIGIBILITY:
Inclusion Criteria:

1. Acute skin, intestinal (histologically confirmed) or liver GvHD > grade 1 according to standard criteria
2. Age ≥18 years
3. Failure of previous treatment, defined as presence of at least one of the following criteria:

   1. Treatment with prednisone/prednisolone/methylprednisolone in a dose of at least 2 mg/kg and lack of response after at least 7 days treatment
   2. Treatment with prednisone/prednisolone/methylprednisolone in a dose of at least 2 mg/kg and progression after at least 3 days of treatment
   3. Failure to taper the prednisone/prednisolone dose to <0.6 mg/kg/day or methylprednisolone dose to <0.5 mg/kg/day
4. Written informed consent
5. Ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

1. Uncontrolled underlying disease
2. Active bleeding
3. Absence of clinical signs of acute GvHD
4. Diagnostic or distinctive clinical signs of chronic GvHD
5. Uncontrolled bacterial, viral or fungal infection
6. Absolute neutrophil count <0.5x103/µl
7. Evidence of transplant-associated micrioangiopathy (TAM) (According to Jodele et al., 2015, diagnostic criteria for TAM)
8. Any previous JAK2 inhibitor treatment prior to study enrolment, except Ruxolitinib given prior to the allogeneic stem cell transplantation
9. Known Hypersensitivity to Ruxolitinib or any of the excipients
10. Known positivity for HIV, Hepatitis B or Hepatitis C at the time of screening.
11. Female patients who are pregnant or breast feeding
12. Concomitant use of any other investigational drug within the last thirty days before the start of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
efficacy of Ruxolitinib and BAT as compared to BAT alone at day 28 after randomisation | at day 28 after randomisation
  To evaluate efficacy of Ruxolitinib and BAT as compared to BAT alone at day 28 after randomisation start in steroid-refractory acute GvHD, measured as response rate

CONTACTS AND LOCATIONS:
Overall Officials: Nikolas von Bubnoff, Professor, Principal Investigator — Medical Center - University of Freiburg
Locations (11):
- Germany (11):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Dresden, Dresden
  - University Medical Center, Freiburg im Breisgau
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Marburg, Marburg
  - Universitätsklinikum München TU rechts der Isar, München
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Bubnoff N, Ihorst G, Grishina O, Rothling N, Bertz H, Duyster J, Finke J, Zeiser R. Ruxolitinib in GvHD (RIG) study: a multicenter, randomized phase 2 trial to determine the response rate of Ruxolitinib and best available treatment (BAT) versus BAT in steroid-refractory acute graft-versus-host disease (aGvHD) (NCT02396628). BMC Cancer. 2018 Nov 19;18(1):1132. doi: 10.1186/s12885-018-5045-7. PMID 30453910
- See also: BMC Cancer. 2018 Nov 19;18(1):1132. doi: 10.1186/s12885-018-5045-7 — https://doi.org/10.1186/s12885-018-5045-7